CLINICAL TRIAL: NCT02433587
Title: Evaluation of Short Versus Long Duration Dual Antiplatelet Therapy in Patients Undergoing Lower Extremity Endovascular Revascularization
Brief Title: Short vs Long Duration Dual Antiplatelet Therapy in Patients Undergoing Lower Extremity Endovascular Revascularization
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Never recruited any patients.
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Vikram S. Kashyap, M.D., Chief, Division of Vascular Surgery & Endovascular Therapy, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-14-29
Record Dates: First submitted 2015-04-29; First posted 2015-05-05 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Peripheral Arterial Disease; Endovascular Procedures
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short Term (Experimental): The short term group will continue Aspirin 81mg and Clopidogrel 75mg for 1 month after the intervention. After that, they will continue Aspirin 81mg only.
  Interventions: Drug: Aspirin; Drug: Clopidogrel
- Long Term (Experimental): The long term group will continue Aspirin 81mg and Clopidogrel 75mg for 6 months after the intervention. After this time, they will continue on Aspirin 81mg only.
  Interventions: Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin — Patients will take Aspirin 81 mg
  Other Names: Acetylsalicylic acid (ASA)
Drug: Clopidogrel — Patients will take Clopidogrel 75 mg
  Other Names: Plavix

SUMMARY:
The primary objective of the trial is to evaluate short versus long duration dual antiplatelet therapy in patients undergoing lower extremity endovascular revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent before initiation of any study related procedures
2. Be at least 18 years of age
3. Successful percutaneous lower extremity (iliac and infrainguinal) endovascular revascularization (percutaneous transluminal angioplasty, and /or stent).
4. At least 1 vessel run-off in segment distal to the intervention
5. Rutherford Classification 2-5 that is unresponsive to medical therapy

Exclusion Criteria:

1. Acute limb ischemia
2. Procedure includes device deployment that has specific FDA regulations for anticoagulation/anti-platelet medication regimen.
3. Patient undergoing atherectomy procedure
4. Intervention includes deployment of drug eluted stent
5. Critical limb ischemia (Rutherford Classification 6)
6. Thrombocytopenia: Platelet count <50k
7. Liver disease (Childs-Pugh B or C)
8. Existing need for on going clopidogrel therapy
9. Proton Pump Inhibitor Use (If unable to be switched)
10. Need for therapeutic anticoagulation
11. Known hypercoagulable disorder
12. Allergy or contraindication to aspirin or clopidogrel
13. Pregnancy
14. Patients enrolled in another investigational drug or device study within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Event Rates | 12 months post-intervention
  Stroke, Myocardial Infarction, Cardiovascular Death
Major Adverse Limb Event Rates | 12 months post-intervention
  Severe limb ischemia leading to a reintervention or major vascular amputation

SECONDARY OUTCOMES:
Quality of Life Outcome | 12 Months post-intervention
  Assessed by Intermittent Claudication Questionnaire and Short Form-36 Health Survey

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States